CLINICAL TRIAL: NCT05525429
Title: Integrated Approach to Enhance Milk Consumption by Vulnerable Household Members in Rural Nepal
Brief Title: Enhancing Milk Consumption by Vulnerable Household Members in Rural Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Heifer Project International (Other)
Responsible Party: Principal Investigator, Laurie Miller, MD, Professor of Pediatrics, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00002768
Record Dates: First submitted 2022-05-21; First posted 2022-09-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education (Active Comparator): Households in this arm will participate in a multidimensional nutrition education intervention, including (1) didactic training on family nutrition (mothers, fathers, adolescent girls), (2) participatory learning activities (mothers, fathers, adolescent girls), (3) model kitchens (mothers, adolescent girls), and (4) Nutrition Club (adolescent girls).
  Interventions: Behavioral: Nutrition Education
- Control (No Intervention): No intervention will be provided. After the research period is complete, the Control group will receive all inputs described above, but no data will be collected during this time period.

INTERVENTIONS:
Behavioral: Nutrition Education — Multidimensional nutrition education will be provided.
  Arms: Nutrition Education

SUMMARY:
Diet quality is generally poor in rural Nepal, especially among vulnerable household members. Consumption of milk (and other animal source foods [ASF]) could contribute to improvements in diet quality. However, multiple cultural, structural and economic barriers constrain the inclusion of ASF in the diet in these households, even though most raise dairy animals. This study will

1. characterize these barriers in detail
2. conduct a randomized controlled trial to test a multi-dimensional behavior change intervention designed to increase ASF/milk consumption by young children 6-60 months, adolescent girls 10-15 years, and women of child-bearing age (WCBA).

Matched clusters of villages in Kapilbastu and Nawalparasi districts (Nepal) will be randomized to Intervention or Control status. Household surveys will be conducted at baseline and 12 months later to collect demographic, diet, feeding practices, nutrition knowledge, etc. Fathers and adolescent girls will respond to mini-surveys. Growth parameters of children, adolescent girls, and WCBA will be assessed. The intervention consists of 4 components: 1) didactic training (mothers, fathers, adolescent girls), 2) participatory learning activities (mothers, fathers, adolescent girls), 3) model kitchens (mothers, adolescent girls), and 4) Nutrition Club (adolescent girls).

The primary outcome will be the impact of the intervention on diet, household feeding practices, and nutrition knowledge.

DETAILED DESCRIPTION:
Animal-source-foods (ASF) contains nutrients essential to human health. These nutrients are especially important for vulnerable household members (young children, adolescent girls, women of child-bearing age [WCBA]). 1, 2 In developing countries, milk is generally one of the largest sources and most widely consumed animal-based dietary protein 3

Although livestock farmers are more likely than their counterparts to consume ASF 3-5, paradoxically, families that rely on agriculture and livestock production for their livelihoods are significantly food and nutrition insecure households. This is partly due to use of the income earned from livestock for purposes other than improving household diet diversity and quality, and partly due to inadequate knowledge about the importance of doing so. In addition, household food allocation practices and cultural beliefs and taboos impact ASF consumption by individual family members. ASF consumption in Nepal, for example, is often prioritized for the primary household bread winner (usually an adult male) 6. Thus, multiple cultural, structural and economic barriers converge to limit consumption of ASF by vulnerable household memb8rs.

Many governmental and non-governmental organizations attempt to improve diet quality in rural households via nutrition education in hopes of motivating behavior change among participants. However, results of such programs have been inconsistent and generally disappointing 7-9. Even programs which provide a robust agricultural intervention are not always successful in improving diets or child growth 10, 11. Therefore, the study will define the barriers to household ASF consumption in rural Nepal and introduce a package of solutions to overcome these barriers. The design of the intervention builds on prior formative work 1, 12-20 21, and will be tested in a randomized controlled trial. While young children under 5 years of age remain a strong focus of this work, adolescent girls, WCBA and fathers will also be included in the intervention activities.

This intervention addresses implementation gaps identified in the investigators' prior work and incorporates findings in recent literature regarding the effectiveness of specific behavior change interventions on nutrition outcomes 22. The investigators' previous work demonstrated that barriers to improving child nutrition are not overcome by increased income, nutrition education, or enhanced household milk production. Recent work has highlighted the value of specific components of behavior change programs: (1) demonstrations of how to perform the behavior, (2) cooking/recipe demonstrations, (3) restructuring the social environment (e.g., women's groups) and engaging with fathers and other groups not typically included, (4) providing households with prompts/cues, (5) action planning, goal-setting and problem-solving, (6) providing information about health consequences, (7) offering strategies to families to self-monitor behaviors. This planned multi-faceted intervention incorporates these elements to augment the effectiveness of behavior change messaging provided to household members, while strengthening community involvement, fostering sustainability and facilitating scaling-up activities.

ELIGIBILITY:
Inclusion Criteria:

* Households involved with Heifer Project International activities. Mothers participate in women's self-help group. Household has at least 1 child 6-60 months at baseline. Household is will to participate.

Exclusion Criteria:

* unwillingness to participate in the research activity, plans to leave the area within the next 12 months, or child 6-60 months or adolescent girl with physical or other special needs that prevent the ingestion of a normal diet-for-age. For adolescent girls, an additional exclusion criterion is the presence of any issues that interfere with their ability to respond.

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1873 (Actual)
Dates: Start 2024-06-08 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Number of Animal Source Foods Consumed in prior 24 hours (diet recall survey), baseline to endline | ~1 year
  Impact of nutrition education on diet of mothers, children 6-60 months, and adolescent girls will compared between baseline and endline.

SECONDARY OUTCOMES:
Change in height-for-age z score from baseline to endline for children 6-60 months | ~1 year
  Child height in centimeters will be measured at baseline and endline. Results will be converted to z scores using World Health Organization standards. Changes in height-for-age z score between baseline and endline will be compared, and related to child consumption of animal source foods.
Change in head circumference-for-age z score from baseline to endline for children 6-60 months | ~1 year
  Child head circumference in centimeters will be measured at baseline and endline. Results will be converted to z scores using World Health Organization standards. Changes in head circumference-for-age z score between baseline and endline will be compared, and related to child consumption of animal source foods.
Change in BMI from baseline to endline for adolescent girls | ~1 year
  Height in centimeters and weight in kilograms will be measured in adolescent girls 10-15 years of age at baseline and endline. Results will be converted to BMI (kg/m^2) using World Health Organization standards. Changes in BMI between baseline and endline will be compared, and related to adolescent consumption of animal source foods.

CONTACTS AND LOCATIONS:
Locations (1):
- Heifer Project International Nepal, Kathmandu, Nepal, Nepal